CLINICAL TRIAL: NCT06531135
Title: A Randomized Controlled Trial of Psychosocial Interventions Facilitating Positive Psychological Adaptation in Patients With Breast Cancer
Brief Title: A RCT of Psychosocial Interventions Facilitating Positive Psychological Adaptation in Breast Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Koo Foundation Sun Yat-Sen Cancer Center (Other)
Collaborators: Soochow university taipei (Unknown)
Responsible Party: Principal Investigator, Chihtao Cheng, Director, Psychiatric department, KFSYSCC, Taiwan, Koo Foundation Sun Yat-Sen Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210628A
Record Dates: First submitted 2024-07-28; First posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer Female
MeSH Terms: interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- stress management (Experimental): 10 weeks of group intervention of Taiwanese version stress management intervention.
  Interventions: Behavioral: T-CBSM
- Support group (Active Comparator): 5 weeks of supportive group intervention.
  Interventions: Behavioral: Support group

INTERVENTIONS:
Behavioral: T-CBSM — A 10-week remotely-delivered group, lasting about 120 minutes each session.
  Other Names: stress management
  Arms: stress management
Behavioral: Support group — Participants will receive weekly supportive-expressive group intervention for two hours per week for five weeks total.
  Other Names: Supportive-Expressive Group
  Arms: Support group

SUMMARY:
To test the effects of a 10-wk stress management interventions vs. a 5-wk control condition on positive psychosocial adaptation in women being treated for breast cancer. Participants assigned to either of the stress management groups will show better positive psychosocial adaptation compared to those in the control group.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 70 years
* Newly diagnosed breast cancer patients in stages I, II, or III (with no prior history of cancer)
* Literate, without significant cognitive impairments
* Capable of writing and expressing themselves in Chinese

Exclusion Criteria:

* Major psychiatric disorders (such as schizophrenia), personality disorders, and substance addiction (excluding smoking)
* Currently participating in other breast cancer-related psychotherapy studies

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2021-11-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
posttraumatic growth by the PTGI | Baseline (T1), post-intervention (T2), 6 months post-intervention (T3)
  the PTGI a 21-item questionnaire each scored on a range of 0-5.
Distress by the HADS | Baseline (T1), post-intervention (T2), 6 months post-intervention (T3)
  The HADS is a 14-item scale, with seven items relating to anxiety and seven relating to depression. Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression.

SECONDARY OUTCOMES:
Positive and Negative affect | Baseline (T1), post-intervention (T2), 6 months post-intervention (T3)
  The Affect Balance Scale includes 20 adjectives assessing negative and positive mood. Possible scores range from 1-5.
Perceived Stress Management Abilities | Baseline (T1), post-intervention (T2), 6 months post-intervention (T3)
  The Measure of Current Status questionnaire and self-designed items were used to measure abilities learned from the group interventions.
Quality of Life by the SF-36 | Baseline (T1), post-intervention (T2), 6 months post-intervention (T3)
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Wei TIng Wang, Principal Investigator — Soochow University ITaipei)
Locations (1):
- Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Taiwan